CLINICAL TRIAL: NCT01433965
Title: Phase I Trial of Maintenance Lenalidomide in Patients With Acute Myeloid Leukemia or High Risk Myelodysplastic Syndrome Post Allogeneic Bone Marrow Transplantation
Brief Title: Study of Lenalidomide in Patients With Acute Myeloid Leukemia or High Risk Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Celgene (Industry)
Responsible Party: Principal Investigator, Mehrdad Abedi, MD, Professor, University of California, Davis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 230510; UCDCC#227 (Other: UC Davis)
Record Dates: First submitted 2011-09-12; First posted 2011-09-14 (Estimated); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
Keywords: Bone marrow transplantation; Maintenance lenalidomide
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phase I Dose Escalation (Experimental): Subjects are given a single dose of the drug while they are observed and tested for a period of time. If they do not exhibit any adverse side effects the dose is escalated, and a new group of subjects is then given a higher dose.
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide will be taken orally once a day for 21 days continuously in 28 day cycles. The dose of the lenalidomide administered to each patient will be based on the group that the patient is enrolled. The dose cycles will be 21 days of a 28 day cycle.
  Other Names: REVLIMID; CC-5013

SUMMARY:
The purpose of this study is to determine whether lenalidomide can stop the growth of leukemia stem cells and can be used to prevent the return of leukemia cells after a transplant.

DETAILED DESCRIPTION:
The purpose of this study is determine whether lenalidomide can directly inhibit leukemic stem cells in vivo and can be used to prevent the relapse of leukemia stem cells after transplant. A concern with any post transplant intervention is the possibility of multiple drug interactions, potential for graft versus host disease exacerbation and/or induction of cytopenia. Therefore, the smallest doses of lenalidomide (5 mg) that has been used in this setting will be utilized as dose level 1. Starting six months post-transplant, patients will begin on a daily dose of lenalidomide. Dependent on the cohort, patients will receive 5 to 20 mg of lenalidomide post transplant. The maximum tolerated dose (MTD) will be determined by the incidence of grade III-IV toxicities of all organs and grade II-IV GVHD. Duration of treatment is six months.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form
* Age greater than or equal to 18 and less than or equal to 65 years
* Able to adhere to the study visit schedule and other protocol requirements.
* High risk acute myelogenous leukemia or high risk myelodysplastic syndrome status post allogeneic bone marrow transplant
* ECOG performance status of less than or equal to 2
* Disease free of other malignancies beside the AML or MDS for ≥ 2 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast.
* All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days and again within 24 hours prior to prescribing lenalidomide for Cycle 1 (prescriptions must be filled within 7 days as required by RevAssist) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy.
* Between 6 months to 8 months post transplant
* Laboratory tests:
* Neutrophil count of ≥ 1.5 x 109/L
* Platelet count ≥ 50 x 109/L
* Calculated creatinine clearance ≥ 60ml/min by Cockcroft-Gault formula
* Total bilirubin ≤1.5 x upper limit of normal
* AST (SGOT) and ALT (SGPT) ≤ 3 x upper limit of normal

Patients are eligible to start on this protocol if they are between 6 months to 10 months post transplant.

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
* Pregnant or breast feeding females (Lactating females must agree not to breast feed while taking lenalidomide)
* Any level of acute graft versus host disease
* Active, uncontrolled infection are not eligible for this study
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Use of any other experimental drug or therapy within 28 days of baseline.
* Known hypersensitivity to thalidomide
* Development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drug
* Known sero-positive for active viral infection with HI, hepatitis B virus (HBV) or hepatitis C virus (HCV)
* Mixed chimerism (at 6 months post transplant will not be started on the protocol
* Active AML or MDS at the time of the study are not eligible for this protocol
* Not able to swallow the lenalidomide capsule as a whole are excluded from this study
* Impaired gastrointestinal absorption

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-08-08 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2021-01-12 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose as assessed by NCI CTCAE, Version 4.0 and Graft versus Host Disease Staging | 4 week cycle; the expected time frame is 24 weeks (or 6 cycles)
  All patients will be followed closely and evaluated for toxicity. For grade III-IV non hematological toxicity or grade IV hematological toxicity associated with lenalidomide will be held until the toxicity resolves and then will be started at a lower dose; Patients who develop grade II to IV GVHD on study will stop lenalidomide

SECONDARY OUTCOMES:
Disease relapse | One year
  Percentage of patients with relapse from all the patients who received the transplant.
Disease-free survival | One year
  Percentage of patients who are alive and remain in remission at one year after infusion of stem cells
Incidence of Graft versus Host disease | One year
  The percentage of pathologically confirmed cases of acute and/or chronic Graft versus Host disease at one year post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Mehrdad Abedi, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis, Sacramento, California, United States